CLINICAL TRIAL: NCT05817006
Title: Early Diagnosis, Prognosis and Prevention of Postcovid Syndrome in Children During the Pandemic of the New Coronavirus Infection COVID-19
Brief Title: Research of the Long-COVID-19 Syndrome in the Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: qwe123456789$
Record Dates: First submitted 2023-02-09; First posted 2023-04-18 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: laboratory and physical examination of postcovid syndrome in children aged 6 to 18 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-COVID-19 (Experimental): conducting laboratory tests, questionnaires, physical examination
  Interventions: Genetic: Device

INTERVENTIONS:
Genetic: Device — research of the long-COVID-19 in the children

SUMMARY:
During the pandemic of the new coronavirus infection COVID-19 in the world community, in the Russian Federation, in particular in the Samara region throughout the pandemic period from the end of 2019, when the first outbreak of a new coronavirus infection occurred in Wuhan (Hubei Province) in the People's Republic of China, the main focus on prevention (development of modern vaccines), diagnosis, treatment and further rehabilitation was done on the adult population. Children acted mainly as carriers of this infection and the manifestation of the disease usually occurred in most cases (not counting children with comorbid conditions) in a mild or latent form. At the moment, after 2 years, we can say that postcovid syndrome also occurs in children, regardless of the severity of the disease.

DETAILED DESCRIPTION:
. During the pandemic of the new coronavirus infection COVID-19 in the world community, in the Russian Federation, in particular in the Samara region throughout the pandemic period from the end of 2019, when the first outbreak of a new coronavirus infection occurred in Wuhan (Hubei Province) in the People's Republic of China, the main focus on prevention (development of modern vaccines), diagnosis, treatment and further rehabilitation was done on the adult population. Children acted mainly as carriers of this infection and the manifestation of the disease usually occurred in most cases (not counting children with comorbid conditions) in a mild or latent form. At the moment, after 2 years, we can say that postcovid syndrome also occurs in children, regardless of the severity of the disease.

Post-COVID syndrome (Post-COVID syndrome, Long COVID) is a long-term symptoms lasting 12 or more weeks. In most cases, it manifests itself as a disorder of autonomic and psychological functions (cognitive impairment), to a lesser extent somatic disorders, prolonged subfebrility.

If you look at the world statistics, according to the World Health Organization, from December 2019 to October 2021, the number of sick children was:

* from 0 to 5 years (children under one year and younger) - 1,890,756, which is only 2% of all reported cases of COVID-19 in the entire world community. The mortality rate in this group of children was 1,797, or 0.1% of the registered deaths worldwide.
* from 5 to 14 years old (older children) - 7,058,748, the indicator has slightly increased and accounts for 7% of all reported cases of COVID-19 in the entire world community. The mortality rate in this group of children is slightly lower, amounting to 1,328, or, as in the previous group, 0.1% of the registered deaths worldwide.
* from 15 to 24 years old (older adolescents and young people, as there is a different age group in the world community) - 14,819,320, which is 15% of all reported cases of COVID-19 in the world. Mortality in this group is 7,023, or 0.4% of all registered deaths in the world. The total mortality among children, adolescents and young people aged 0 to 25 years was less than 0.5% of the registered deaths in the world.

Worldwide, and in the Russian Federation in particular, in 2022, the incidence of COVID-19, according to WHO, among children has increased sharply against the background of an increase in the incidence of the Omicron strain at a time when most countries have weakened public health and social measures. For example, in the United States, by July 2022, there were 14,003,497 cases of the disease in children, and the children were 18,6% (14 003 497 /75 463 921) of all registered cases, with a total of 18,605 cases per 100,000 children in the population. Worldwide, by July 24, 2022, the proportion of children under the age of 5 and children aged 5 to 14 years was 2.47% and 10.44%, respectively. Adolescents and young people aged 15 to 24 accounted for 13.91% of all cases. Children aged 5 years and younger account for 0.11% of all deaths in the world, while children aged 5 to 14 years account for 0.089%, and adolescents and young people account for 0.37% of all reported deaths in the world.

In the Russian Federation, there are no statistics on the incidence of a new coronavirus infection in children, there are separate data by region, but there are no general statistics. In this regard, it can be assumed that a large number of children who have suffered COVID-19 is not taken into account, so it is necessary to investigate the postcovid syndrome not only in children who have suffered a new coronavirus infection with confirmed laboratory data, but also in those who have suffered it asymptomatically or under the guise of a common respiratory infection in order to identify long-term and chronic symptoms COVID-19 in children. Having studied the main biological mechanisms that cause these symptoms, researchers will be able to identify patients at risk of chronic infection, prevent the development of such conditions and will be able to carry out early rehabilitation of children who have suffered COVID-19.

ELIGIBILITY:
Inclusion Criteria:

• children from 6 to 18 years

Exclusion Criteria:

• no

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-16 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
postcovid syndrome in children | 1 year
  Number of Participants with research of the bridge syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Olga Borisova, Study Director — Doctor of Sciences, Professor
Locations (1):
- Danija, Samara, Pestravka, Russia

IPD SHARING:
Plan to Share IPD: Yes
development of a unified integrated model for assessing neurological status, cognitive disorders, somatic disorders of organs and systems to identify patients at risk of chronic infection, prevent the development of such conditions, conduct early personal rehabilitation of children who have undergone COVID-19, and further develop methods for conducting medical examinations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: available to everyone